CLINICAL TRIAL: NCT06367400
Title: Validation of Pediatric Sleep Questionnaire, a Multi-center Study in Sweden
Brief Title: Validation of Pediatric Sleep Questionnaire on a Swedish Cohort
Status: Recruiting | Type: Observational
Sponsor: Uppsala University (Other)
Collaborators: Karolinska Institutet (Other); Örebro University, Sweden (Other); Umeå University (Other); Göteborg University (Other)
Responsible Party: Sponsor
Other Study IDs: SwePSQ
Record Dates: First submitted 2024-04-03; First posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Obstructive Sleep Apnea; Sleep Disorder; Sleep Disorders in Children; Obstructive Sleep Apnea of Child
Keywords: OSDB; PSQ; Pediatrics
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Wake Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PSQ-cohort: Patients recruited from Akademiska Sjukhuset, Örebro, Västra Götaland, Skåne, Stockholm and Umeå.
  Interventions: Diagnostic Test: Pediatric Sleep Questionnaire

INTERVENTIONS:
Diagnostic Test: Pediatric Sleep Questionnaire — Questionnaire with 22 questions of symptoms of OSDB

SUMMARY:
This study is aimed to validate the questionnaire called Pediatric Sleep Questionnaire on a Swedish cohort of children from 18 months to 15 years old with obstructive sleep disordered breathing.

ELIGIBILITY:
Inclusion Criteria:

* Children with OSDB-symptoms referred to ENT-clinics
* Age between 18 months and 15 years old.
* Good knowledge of the Swedish language

Exclusion Criteria:

* Craniofacial abnormalities
* Mb Down
* neuromuscular disorders
* do not understand swedish

Ages: 18 Months to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population will be included from the ENT-clinics or the waiting lists to surgical treatments.
Sampling Method: Non-Probability Sample
Enrollment: 520 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2034-12-31 (Estimated)

PRIMARY OUTCOMES:
Level of baseline PSQ | Baseline
  Level of baseline PSQ of children who are referred to surgery. A level of >33% yes i.e. 8/22 indicates medium to severe OSA and less than five yes indicates a healthy status. Minimum is 0 yes and maximum is 22 where 22 is the most severe disease.
  PSQ has a score from 0 to 22 where every yes on the scale is one point. A level of 8 "yes" (>33%) indicates moderate to severe OSDB and less than five indicates no OSDB.
Changes of baseline PSQ after treatment | 6 months to 12 months
  Changes of baseline PSQ with 6 months follow-up, after treatment/surgery

SECONDARY OUTCOMES:
PSQ vs OSA-18 | 6 months
  Compare PSQ-levels with OSA-18 levels OSA-18 is accounted as a scale from 18 to 126 points where a higher rate is a more severe disease. Score less than 60 suggests a mild impact on quality of life. Scores between 60 and 80 a moderate impact and a score higher than 80 severe impact.
  OSA-18 has a summary of 18 - 126 points where a higher level indicates worse quality of life. A score less than 60 indicates a mild impact on quality of life and score between 60 and 80 indicates moderate impact whereas a score above 80 indicates a high impact.
PSQ vs. PSG | 6 months
  PSQ-levels compared to Polysomnography outcomes
PSQ levels of healthy controls vs children with OSDB | 6 months
  Compare the PSQ-levels of children with OSDB-symptoms to children without OSDB-symptoms

OTHER OUTCOMES:
5 and 10 years follow-up | 11 years
  PSQ and OSA-18 compared to baseline and after 6months compared to levels at 5 and 10 years follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Akademiska hospital, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No